CLINICAL TRIAL: NCT00912054
Title: DuoTrav APS Versus XALACOM® in Ocular Surface Health
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-007
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-01

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: OAG; OH
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Xalacom

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): DuoTrav APS
  Interventions: Drug: DuoTrav APS
- 2 (Active Comparator): Xalacom
  Interventions: Drug: Xalacom

INTERVENTIONS:
Drug: DuoTrav APS — travoprost APS 40 micrograms/ml / timolol 5 mg/ml, Eye Drops, Solution, once daily
  Arms: 1
Drug: Xalacom — XALACOM® (latanoprost 50 micrograms/ml / timolol 5 mg/ml) Eye Drops, Solution
  Arms: 2

SUMMARY:
To demonstrate superiority of DuoTrav APS over XALACOM® in Ocular Surface Health in patients with open angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age.
2. Must have a clinical diagnosis of open-angle glaucoma (with or without pseudoexfoliation or pigment dispersion component), or ocular hypertension in at least one eye.
3. Must be willing and able to discontinue use of any topical ocular medication other than the study medication for the duration of the study.
4. Must have had IOP controlled with mono-therapy using XALACOM for at least 1 continuous month prior to Visit 1.
5. Women of childbearing potential must meet all specific conditions at Visit 1:

Exclusion Criteria:

1. Any abnormality preventing reliable applanation tonometry in the study eye(s).
2. Presence of any ocular pathology in either eye seen during the slit lamp or fundus exams that may preclude the safe administration of test article or safe participation in this study.
3. Dry eye or KCS which has been, or is currently being, treated with the use of punctal plugs, punctal cautery, Restasis®, or topical ocular corticosteroids.
4. Patients who have undergone keratorefractive ocular laser procedures, corneal surgery or surgery to the corneal surface, within 1 year prior to Visit1
5. Any other ocular laser surgery in either eye within 3 months
6. Patients who have undergone intraocular or extra-ocular surgery, in either eye, within 6 months prior to Visit 1.
7. History of other progressive retinal or optic nerve disease.
8. Severe central visual field loss in either eye based upon the clinical judgment of the investigator.
9. Any history of, or current evidence of, infectious or inflammatory ocular conditions
10. Ocular trauma within 6 months prior to Visit 1 in either eye, as determined by patient history and/or examination.
11. History or evidence of corneal transplant or transplant variant procedures
12. Patients with suspected or diagnosed Sjogren's syndrome.
13. History of or current bronchial asthma, or severe chronic obstructive pulmonary disease
14. History of or current severe, unstable or uncontrolled cardiovascular, hepatic, or renal disease.
15. History of spontaneous or current hypoglycemia or uncontrolled diabetes.
16. History of or current severe allergic rhinitis and bronchial hyper reactivity.
17. Intolerance/hypersensitivity to any component of the medication
18. Use of any systemic medications on a chronic basis that have not been on a stable dosing regimen for at least 30 days prior to Visit 1, or an anticipated change in dosing regimen of medications during the course of the study.
19. Use of ocular medications other than XALACOM® within 7 days
20. Use of corticosteroids within 30 days of Visit 1, or any anticipated use of corticosteroids during the course of the study.
21. Use of contact lenses within 30 days of Visit 1. Concomitant use of contact lenses is also excluded for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline (Day 0) in Ocular Surface Disease at the end of the treatment period (Day 90) | Visits 1 and 3

SECONDARY OUTCOMES:
Percent of patients with a corneal fluorescein staining score of 0 at the end of the treatment period (Day 90) | Visit 3 (Day 90)

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium